CLINICAL TRIAL: NCT05782803
Title: Investigation of the Effect of Craniocervical Flexion Training on Suprahyoid Muscles in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, ARZUCAN TOKSAL, Lecturer, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: ZonguldakBulentEcevitU
Record Dates: First submitted 2023-03-07; First posted 2023-03-24 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Dysphagia; Rehabilitation; Stability
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercises Group (Experimental): As stated in the literature, 20 sessions of KSF training will be given to the study group for 4 weeks.
  Interventions: Behavioral: Exercises Group
- Control Group (No Intervention): Participants in the control group will not receive intervention throughout the study.

INTERVENTIONS:
Behavioral: Exercises Group — A Pressure Biofeedback Device will be used in CCF training to increase awareness and focus on the desired muscle. After the person is brought to the hook position, the pressurized biofeedback device will be placed in the middle position between the craniocervical and cervical vertebrae or horizontally so that the protrusion between the earlobe and the chin is removed. It is inflated to a standard 20 mmHg to ensure surface-to-longitudinal contact. Participants are taught the correct craniocervical flexion movement without first working the superficial muscles. The patient is then asked to look with their eyes slightly toward the chest cavity. During the exercises, starting from 20 mmHg and increasing by 2 mmHg, the desired level of 30 mmHg will be reached. At each level, the movement is continued for 10 seconds, resting for 3-5 seconds, 10 repetitions are required. If the same level is maintained for 10 seconds and 10 repetitions, the next level is passed.
  Arms: Exercises Group

SUMMARY:
Swallowing; It is a complex, dynamic, sensorimotor process involving more than 30 muscles located bilaterally in the oral, pharyngeal, and esophageal regions and involving the safe delivery of the food taken from the mouth to the stomach as a result of sequential and coordinated movements. The cervical region is important in terms of swallowing function, as it acts as a bridge between the oral and esophageal structures through the pharynx, hosts the larynx and upper respiratory tract, which plays an important role in safe swallowing, and contributes to the stabilization and preservation of posture thanks to the muscles in its structure. Craniocervical flexion (CCF) occurs at the atlantooccipital joint and upper cervical segments such as C1-2. While superficial muscles such as the SCM and anterior scalene muscles contract in cervical flexion, deep muscles such as the longus colli and capitis, which are mainly primary cervical stabilizer muscles, are activated in CCF. CCF is a movement felt as flexion in the upper part of the cervical region with a slight retraction of the chin. It is also known that the suprahyoid muscles are activated in CCF. Swallowing in the CCF posture has been shown to occur with less suprahyoid muscle activation. The cervical region must provide proper alignment, posture, and stabilization for effective and safe swallowing. Postural changes in the cervical region, and changes in the position of the hyoid bone cause changes in gravity, oropharyngeal structures, and muscle length-tension relationship, thereby changing the dynamics of swallowing function. Therefore, it is not possible to consider the cervical region separately from the swallowing function. However, the focus of the exercises to be chosen for the cervical region is different and the effects that are likely to occur may also be different. There is no study in the literature on the activation of superficial and deep muscles activated during swallowing of craniocervical flexion training exercises, which aim to improve cervical region mechanics by focusing especially on deep cervical flexors. The aim of this study is to investigate the effect of craniocervical flexion training (CCF) on swallowing-related structures in healthy individuals.

DETAILED DESCRIPTION:
Swallowing; It is a complex, dynamic, sensorimotor process involving more than 30 muscles bilaterally located in the oral, pharyngeal, and esophageal regions, and involving the safe delivery of food taken from the mouth to the stomach as a result of sequential and coordinated movements. The cervical region is important in terms of swallowing function as it acts as a bridge between the mouth and esophagus structures through the pharynx, contains the larynx and upper respiratory tract, which plays an important role in safe swallowing, and contributes to stabilization. Maintaining posture thanks to the muscles in their structure. Craniocervical flexion (CCF) occurs at the atlantooccipital joint and upper cervical segments such as C1-2. In cervical flexion, the superficial muscles such as the SCM and anterior scalene muscles contract, whereas in CCF, mainly deep muscles such as the longus colli and capitis, which are the primary cervical stabilizer muscles, are activated. CCF is a movement felt as flexion in the upper part of the cervical region with slight retraction of the chin. It is also known that the suprahyoid muscles are activated in CCF. It has been shown that swallowing in the CCF stance occurs with less suprahyoid muscle activation. For effective and safe swallowing, the cervical region must provide proper alignment, posture, and stabilization. Postural changes in the cervical region and changes in the position of the hyoid bone cause changes in gravity, oropharyngeal structures, and muscle length-tension relationship, thereby changing the dynamics of swallowing function. Therefore, it is not possible to consider the cervical region separately from the swallowing function. However, as the focus of the exercises to be chosen for the cervical region is different, the possible effects may also be different. There are no studies in the literature on the activation of superficial and deep muscles activated during swallowing of craniocervical flexion training exercises, which aim to improve cervical region mechanics, especially by focusing on deep cervical flexors. The aim of this study is to investigate the effect of craniocervical flexion training (CCF) on swallowing structures in healthy individuals. At least 50 people meeting the inclusion criteria of Zonguldak Bülent Ecevit University will be included in the study and will be equally divided into groups by randomization. After the individuals included in the study have read and accepted the informed consent form, the following evaluations will be applied first. Evaluations begin with filling out the demographic data form, cervical region normal joint range of motion, cervical region muscle strength, cervical region posture analysis, craniocervical flexion test, activity score and performance value of deep cervical flexor muscles, evaluation of suprahyoid muscles by superficial EMG evaluation method, water drinking test Evaluation of swallowing function will be done with Assessments will take 25-30 minutes. After the initial evaluations, the participants will be randomized by the closed envelope method and divided into the exercise group and the control group. As stated in the literature, 20 sessions of KSF training will be given to the study group for 4 weeks. No intervention will be made to the control group during this period. After the exercise sessions are completed, the same evaluations will be repeated for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old and volunteering.
* Having a Mini-Mental test score of 24 and above

Exclusion Criteria:

* Having a history of cervical trauma, cervical disc herniation, and osteoarthritis
* Having a history of additional disease that interferes with assessments and physical activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Surface Electromyographic Measurements of the Suprahyoid Muscles | 4 months
  yEMG, which provides practical objective data and provides electrical activation information directly from the relevant muscles, will measure the activation development in the muscles during the maximum voluntary isometric contractions to be made during a standard activity (drinking 10 ml of water). The EMG measurement to be applied to the participants will be done outside working hours in a way that will not disrupt routine patient functioning. The electrodes to be used in EMG will be covered by the researchers. This assessment will be applied before the start of the exercise program and at the end of the exercise program at the end of the 4th week.

SECONDARY OUTCOMES:
Evaluation of Normal Joint Range of Motion of the Cervical Region | 4 months
  The range of motion of the cervical region (flexion, extension, right and left lateral flexion, right and left rotation) will be evaluated by the goniometer, as indicated in the literature, by placing the patient in a suitable position in a quiet and calm environment. The measurement will be repeated 3 times and the average values will be taken.
Evaluation of Cervical Region Muscle Strength | 4 months
  Cervical flexion, cervical extension, cervical right and left lateral flexion, cervical right and left rotation will be evaluated by manual muscle test, by giving the patient an appropriate position in an appropriate environment.
Cervical Posture Analysis | 4 months
  Anterior and lateral cervical postural analysis will be performed. In the anterior posture analysis, deviation to the right or left according to the relationship between the chin and the suprasternal pit and the height difference of both shoulders will be evaluated with the anterior gaze. In the lateral posture analysis, protraction and retraction of the shoulders with forward or backward deviation will be evaluated according to the shoulder joint vertex-auricle relationship with the lateral gaze.
Craniocervical Flexion Test (CCFT) | 4 months
  the uninflated pressure sensor (Stabilizer, Chattanooga, USA) is placed between the projection of the earlobe and the chin and inflated to the initial pressure of 20 mmHg. This is standard pressure that is sufficient to fill the gap between the neck and the surface to be tested but will not increase lordosis. The instrument provides feedback and guidance to the patient to perform the five phases required for testing. The movement is done lightly and slowly as if to nod the head (as if to say yes). The CSFT will be used to test the activation and endurance of the deep neck flexors in progressive increments of 2 mmHg from 20 mmHg to 30 mmHg, maintaining isometric contractions at progressive pressures.

CONTACTS AND LOCATIONS:
Overall Officials: Arzucan Toksal, Phd Candidate, Study Director — Zonguldak Bulent Ecevit University
Locations (1):
- Zonguldak Bülent Ecevit University, Zonguldak, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jull GA, O'Leary SP, Falla DL. Clinical assessment of the deep cervical flexor muscles: the craniocervical flexion test. J Manipulative Physiol Ther. 2008 Sep;31(7):525-33. doi: 10.1016/j.jmpt.2008.08.003. PMID 18804003
- [Background] Kilinc HE, Unver B. Effects of Craniocervical Flexion on Suprahyoid and Sternocleidomastoid Muscle Activation in Different Exercises. Dysphagia. 2022 Dec;37(6):1851-1857. doi: 10.1007/s00455-022-10453-1. Epub 2022 Apr 26. PMID 35471669